CLINICAL TRIAL: NCT06554483
Title: The Effects of Neuroscience Based Proprioceptive Exercise Training in Elderly With Chronic Knee Pain
Brief Title: The Effects of Neuroscience Based Proprioceptive Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fatih Tekin, Assist. Prof., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NEUROSCIENCE IN KNEE PAIN
Record Dates: First submitted 2024-07-25; First posted 2024-08-15 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Chronic Knee Pain; Pain, Chronic; Elderly
MeSH Terms: conditions — Chronic Pain | interventions — Exercise; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: The participants will assigned to the experimental or control group by randomization method. Each group will include in an exercise program for 6 weeks, 2 sessions per week, each session for an average of 60 minutes. The exercise program of the experimental group consist of a combination of a 10-minute warm-up period with graded walking, mobility and stretching exercises, a 20-minute proprioceptive exercise program, a 20-minute nbpet using a laser pointer, and stretching and relaxation exercises that ended with a 10-minute cool-down period. Control group's exercise program consist of a 10-minute warm-up period with graded walking, mobility and stretching exercises, followed by a 40-minute proprioceptive exercise program and a 10-minute cool-down period consisting of stretching and relaxation exercises.
Who Masked: Participant
Masking Description: participants will not be informed whether they are in the experimental or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neuroscience based proprioceptive exercise training group (Experimental): Neuroscience based proprioceptive training using laser pointer A pre-created wallpaper indicating various directions is fixed on the wall 90 cm away from the patient (at the level of the patient's knee when the patient is standing upright). Then, the laser pointer (producted by NMC training system) will fixed to the patient's knee with the help of a velcro so as not to interfere with the patient's knee movement. At the beginning of the exercise, the patient is asked to move the light on the laser pointer to the midpoint of the wallpaper. The patient is then asked to follow the instructions on the wallpaper by moving the knee in flexion-extension, medio-lateral directions. These instructions are continued throughout the exercise in different directions. Meanwhile, the patient is asked to perform mild cognitive tasks such as counting numbers, names of people starting with any letter, city names or animal names. The training continued for approximately 20 minutes.
  Interventions: Other: Exercise
- Proprioceptive exercise group (Active Comparator): A proprioceptive training regimen will established with Swiss balls. The proprioceptive activities are advanced on a weekly basis in order to test the patient's balance in response. Patients have training in three stages: beginning, intermediate, and advanced. Each exercise is performed as 3x10 repetitions. Between sets, 2-3 minutes rest breaks is given. The beginning phase is applied in the 1st and 2nd weeks, the intemediate phase in the 3rd and 4th weeks, and the advanced phase in the 5th and 6th weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — supportive reliable exercise programs
  Other Names: Proprioceptive exercise

SUMMARY:
Neuroscience based proprioceptive exercise trainig using laser pointer (nbpet) is a new aproach exercise training method. In this study, This study aimed to investigate the effects of nbpet using laser pointer on different fonctional parameters.

DETAILED DESCRIPTION:
This study aim to investigate the effects of nbpet using laser pointer on different fonctional parameters.

Participants will divide into two groups (experimental and control ). Joint position errors will evaluate with the jonit position error assessment method, range of motion with a goniometer, kinesiophobia with the Tampa kinesiophobia scale, pain with the Mc Gill pain scale, quality of life with the Older People Quality of Life questionnaire (OPQoL-brief), and mobility with the time up and go test. Both groups will include in the exercise program with proprioceptive exercise training for 2 sessions per week for 6 weeks. In addition, the experimental group will train with nbpet using laser pointer at the same time.

Properioceptive training A proprioceptive training regimen will establish with Swiss balls. The proprioceptive activities is advanced on a weekly basis in order to test the patient's balance in response. Patients have training in three stages: beginning, intermediate, and advanced. Each exercise will perform as 3x10 repetitions. Between sets, 2-3 minutes rest breaks will given. The beginning phase will applied in the 1st and 2nd weeks, the intemediate phase in the 3rd and 4th weeks, and the advanced phase in the 5th and 6th weeks. The proprioceptive rehabilitation protocol is based on a previous study. All the program will conducted by one experienced physiotherapist.

Neuroscience based proprioceptive training using laser pointer A pre-created wallpaper indicating various directions will fix on the wall 90 cm away from the patient (at the level of the patient's knee when the patient was standing upright) . Then, the laser pointer (producted by NMC training system) will fix to the patient's knee with the help of a velcro so as not to interfere with the patient's knee movement.

At the beginning of the exercise, the patient is asked to move the light on the laser pointer to the midpoint of the wallpaper. The patient is then asked to follow the instructions on the wallpaper by moving the knee in flexion-extension, medio-lateral directions. These instructions are continued throughout the exercise in different directions. Meanwhile, the patient is asked to perform mild cognitive tasks such as counting numbers, names of people starting with any letter, city names or animal names. The training continues for approximately 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* having a history of knee pain for 6 months or longer
* having unilateral knee pain, being 60 years of age or older, and completing the assessments.

Exclusion Criteria:

* being under 60 years of age, having bilateral knee pain
* being diagnosed with a disease that may cause knee pain (osteatritis, meniscus rupture, ACL rupture...)
* having knee pain for less than 6 months
* have visual and hearing impairments that affect exercise, having knee extension limitations.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
pain meausere | 6 weeks
  Short-form McGill Pain Questionnaire (SF-MPQ) will used to examine pain level of participants. The main component of the SF-MPQ consists of 15 descriptive adjectives for the pain sensation (11 sensory and 4 affective), which are self-rated by the patient according to their intensity level on a point rating scale (0 = none,1 = mild, 2 = moderate, 3 = severe). Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors. The total score is the sum of the intensity values.
position error | 6 weeks
  Joint Position Error measurement will used to asses knee proprioception of elderly. It is a test performed with a wall-mounted board consisting of circles drawn at a distance of 1 cm from the patient and a laser placed on the patient's knee with appropriate belts. After the laser is placed on the patient's knee, the patient stands and tries to hold the laser light at the starting point with eyes open on the board placed 90 cm away. The patient is first asked to perform 10 repetitions of knee flexion and extension and then to return the laser to the starting position with eyes closed. In the final stage, the patient's horizontal, vertical and global distance from the laser light starting point is recorded in cm

SECONDARY OUTCOMES:
Range of motion | 6 weeks
  Knee range of motion assesment: Knee range of motion (KROM) will assesed using a standard goniometer, consisting of a protractor body with two arms (one stationary and one movable), was used for all measurements. Participants are positioned supine on a flat examination table For knee flexion measurements, participants are instructed to lie supine with the hip of the leg being measured in a neutral position. The fulcrum of the goniometer is placed over the lateral epicondyle of the femur, the stationary arm is aligned with the greater trochanter of the femur, and the movable arm is aligned with the lateral malleolus of the fibula
Qualitiy of life | 6 weeks
  Older People Quality of Life questionnaire (OPQoL-brief): OPQoL-brief will used to evaulate quality of life. A shortened version of OPQoL-brief was developed by Bowling et al. The OPQoL-brief consisted of 13 statements, with the participants being asked to indicate the extent to which they agree with each statement by selecting one of five possible options ("strongly disagree," "disagree," "neither agree nor disagree," "agree," and "strongly agree"). The range in the original version is based on the principle of point allocation. The items are summed to provide a total OPQoL-brief score. The total score of OPQoL-brief ranges from 13 to 65 and higher scores indicate better QoL. Te OPQoL - brief questionnaire also includes a preliminary single item on global OoL. This single item is not scored with the OPQOL; it is coded as very good (5) to very bad
Kinesiophobia | 6 weeks
  Tampa Scale for Kinesiophobia (TSK): The TSK-11 will used to asses kinesiophobia. This scale consists of 11 questions. A 4-point Likert scale assigns a score to each item, which includes strongly disagree, disagree, agree, and strongly agree options. The total score ranges from 11 to 44. A high score indicates a high level of kinesiophobia. Individuals were asked to tick the appropriate box for each question, and the total score was calculated.The lowest score on this scale is 11 and the highest score is 44. The higher the score, the higher the kinesiophobia.
Time up and Go test | 6 weeks
  The Time up and Go test (TUG): The TUG will used to evaluate mobility. The TUG is a balance and gait index which requires the patient to stand up from a chair, walk a 3 m distance, turn, walk back to the chair, and sit down. The time required to complete the task is measured in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Aziz DENGIZ, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takahashi A, Kitamura K, Watanabe Y, Kobayashi R, Saito T, Takachi R, Kabasawa K, Oshiki R, Tsugane S, Iki M, Sasaki A, Yamazaki O, Nakamura K. Epidemiological profiles of chronic low back and knee pain in middle-aged and elderly Japanese from the Murakami cohort. J Pain Res. 2018 Dec 12;11:3161-3169. doi: 10.2147/JPR.S184746. eCollection 2018. PMID 30588068
- [Background] Mitchell HL, Hurley MV. Management of chronic knee pain: a survey of patient preferences and treatment received. BMC Musculoskelet Disord. 2008 Sep 18;9:123. doi: 10.1186/1471-2474-9-123. PMID 18801169
- [Background] Bjordal JM, Ljunggren AE, Klovning A, Slordal L. Non-steroidal anti-inflammatory drugs, including cyclo-oxygenase-2 inhibitors, in osteoarthritic knee pain: meta-analysis of randomised placebo controlled trials. BMJ. 2004 Dec 4;329(7478):1317. doi: 10.1136/bmj.38273.626655.63. Epub 2004 Nov 23. PMID 15561731
- [Background] Gutthann SP, Garcia Rodriguez LA, Raiford DS. Individual nonsteroidal antiinflammatory drugs and other risk factors for upper gastrointestinal bleeding and perforation. Epidemiology. 1997 Jan;8(1):18-24. doi: 10.1097/00001648-199701000-00003. PMID 9116088
- [Background] Juni P, Reichenbach S, Egger M. COX 2 inhibitors, traditional NSAIDs, and the heart. BMJ. 2005 Jun 11;330(7504):1342-3. doi: 10.1136/bmj.330.7504.1342. No abstract available. PMID 15947376
- [Background] Beswick AD, Wylde V, Gooberman-Hill R, Blom A, Dieppe P. What proportion of patients report long-term pain after total hip or knee replacement for osteoarthritis? A systematic review of prospective studies in unselected patients. BMJ Open. 2012 Feb 22;2(1):e000435. doi: 10.1136/bmjopen-2011-000435. Print 2012. PMID 22357571
- [Background] Jiang L, Zhang L, Huang W, Zeng Q, Huang G. The effect of proprioception training on knee kinematics after anterior cruciate ligament reconstruction: A randomized control trial. J Back Musculoskelet Rehabil. 2022;35(5):1085-1095. doi: 10.3233/BMR-210201. PMID 35213344
- [Background] Hajouj E, Hadian MR, Mir SM, Talebian S, Ghazi S. Effects of Innovative Aquatic Proprioceptive Training on Knee Proprioception in Athletes with Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial. Arch Bone Jt Surg. 2021 Sep;9(5):519-526. doi: 10.22038/abjs.2020.50106.2485. PMID 34692934
- [Background] Genevsky A, Garrett CT, Alexander PP, Vinogradov S. Cognitive training in schizophrenia: a neuroscience-based approach. Dialogues Clin Neurosci. 2010;12(3):416-21. doi: 10.31887/DCNS.2010.12.3/agenevsky. PMID 20954435
- [Background] Kleim JA, Hogg TM, VandenBerg PM, Cooper NR, Bruneau R, Remple M. Cortical synaptogenesis and motor map reorganization occur during late, but not early, phase of motor skill learning. J Neurosci. 2004 Jan 21;24(3):628-33. doi: 10.1523/JNEUROSCI.3440-03.2004. PMID 14736848
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Woby SR, Roach NK, Urmston M, Watson PJ. Psychometric properties of the TSK-11: a shortened version of the Tampa Scale for Kinesiophobia. Pain. 2005 Sep;117(1-2):137-44. doi: 10.1016/j.pain.2005.05.029. PMID 16055269
- [Background] Bowling A, Hankins M, Windle G, Bilotta C, Grant R. A short measure of quality of life in older age: the performance of the brief Older People's Quality of Life questionnaire (OPQOL-brief). Arch Gerontol Geriatr. 2013 Jan-Feb;56(1):181-7. doi: 10.1016/j.archger.2012.08.012. Epub 2012 Sep 19. PMID 22999305
- [Background] Wall JC, Bell C, Campbell S, Davis J. The Timed Get-up-and-Go test revisited: measurement of the component tasks. J Rehabil Res Dev. 2000 Jan-Feb;37(1):109-13. PMID 10847578
- [Result] Sengupta T, Paul B, Banerjee A, Das R, Halder R. Chronic musculoskeletal pain among elderly individuals in a rural area of West Bengal: A mixed-method study. Malays Fam Physician. 2023 Apr 19;18:25. doi: 10.51866/oa.232. eCollection 2023. PMID 37205144